CLINICAL TRIAL: NCT01690182
Title: Effects of Test Meal Volume and Energy Density on Gastric Volumes and Satiety Assessed by MRI
Brief Title: MRI Study of Stomach Volumes and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: F/11/2010
Record Dates: First submitted 2012-09-17; First posted 2012-09-21 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: Gastrointestinal physiology; MRI; gastric volumes; satiety

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Study test meal 1 (Experimental): High volume, high energy density test meal. Volunteers will be given 490 mL of a high energy test meal once in the morning
  Interventions: Dietary Supplement: Study test meal 1
- Study test meal 2 (Experimental): High volume, low energy density test meal. Volunteers will be given 490 mL of a high volume low energy density test meal once in the morning
  Interventions: Dietary Supplement: Study test meal 2
- Study test meal 3 (Experimental): A low volume, high energy test meal. Volunteers will be given 140 mL high energy density test meal once in the morning.
  Interventions: Dietary Supplement: Study test meal 3

INTERVENTIONS:
Dietary Supplement: Study test meal 1 — Volunteers will be fed with a high volume, high energy density test meal.
  Arms: Study test meal 1
Dietary Supplement: Study test meal 2 — Volunteers will be fed with a high volume, low energy density test meal
  Arms: Study test meal 2
Dietary Supplement: Study test meal 3 — Volunteers will be fed with a low volume, high energy density test meal
  Arms: Study test meal 3

SUMMARY:
The GI MRI Research group at the University of Nottingham has been developing new, non-invasive magnetic resonance imaging (MRI) techniques to image the gastrointestinal tract. In collaboration with food manufacturer Unilever, the investigators want to image the abdomen of healthy volunteers after consumption of test meals of varying volume and energy density to determine levels of gastric distension and investigate possible correlations of this with the subjects' sense of satiety.

DETAILED DESCRIPTION:
The tone of the proximal stomach decreases on meal intake through a process of gastric accommodation, aimed at increasing the capacity of the stomach. An increased gastric volume progressively distends the stomach, and this distension has been shown to have an inverse relationship on appetite. The link is assumed to be based on activation of mechanoreceptors lying in the walls of the stomach. On activation, vagal discharges are triggered, leading to activation of hypothalamic neurons and regulation of feelings of satiety. Gasrtric emptying is also regulated by duodenal feedback mechanisms triggered by the arrival and amount of nutrients.

Based on current knowledge, a high volume test meal would be expected to produce more gastric distension and satiety over a low volume test meal, and a low energy density food would be expected to empty from the stomach faster than a high energy density food. Going on this premise, study test meal 2 would be expected to empty faster than study test meal 1. These phenomena will be investigated using non invasive Magnetic Resonance Imaging (MRI) methods. MRI can measure gastric volumes serially and non-invasively with high spatial resolution. Ultimately, the findings from this study will provide novel insights on mechanisms of gastric distension and satiety.

ELIGIBILITY:
Inclusion criteria:

* Apparently healthy; no medical conditions that might affect the study measurements (as determined by the study physician)
* No use of medication that would interfere with the study measurements (as determined by the study physician)
* No use of antibiotics in the 3 months before the study or during the study
* No reported participation in another nutritional or biomedical trial 3 months before the study or during the study
* Being used to eating 3 meals daily
* BMI: 20 - 35 kg m-2
* No reported participation in night shift work 2 weeks prior to the study or during the study
* Not taking part in strenuous exercise ≤10 hours/week
* Not consuming more than 21 alcoholic test meals in a typical week
* Not presently a smoker
* No reported weight loss or gain of more than 10 % of bodyweight for 6 months before the study
* No eating disorder
* No MRI contraindications; i.e absence of metal implants, infusion pumps and pacemakers, as assessed by a MRI safety screening questionnaire

Exclusion criteria:

* High or very high restrained eater
* Use of any medically- or self-prescribed diet for the duration of the study
* Allergies or food intolerances

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Total gastric content half emptying time T50 | 0 - 240 mins
  Total gastric volume at half the experimental time

SECONDARY OUTCOMES:
Volumes of test meal in the stomach | 0 - 240 mins
  gastric volumes of the test meals in the stomach obtained from MRI images, as a function of time

OTHER OUTCOMES:
Relationship of gastric behaviour of test meal stomach volumes with satiety | 0 - 240 minutes
  A comparison of the gastric volumes with satiety scores obtained throughout the experiment

CONTACTS AND LOCATIONS:
Overall Officials: Luca Marciani, PhD, Principal Investigator — University of Nottingham
Locations (2):
- Unilever Research and Development, Olivier Van Noortlann 120, AT Vlaardingen, Netherlands
- Nottingham Digestive Diseases Centre and Sir Peter Mansfield Magnetic Resonance Centre, University of Nottingham, Nottingham, United Kingdom

REFERENCES:
- [Derived] Murray K, Placidi E, Schuring EA, Hoad CL, Koppenol W, Arnaudov LN, Blom WA, Pritchard SE, Stoyanov SD, Gowland PA, Spiller RC, Peters HP, Marciani L. Aerated drinks increase gastric volume and reduce appetite as assessed by MRI: a randomized, balanced, crossover trial. Am J Clin Nutr. 2015 Feb;101(2):270-8. doi: 10.3945/ajcn.114.096974. Epub 2014 Dec 3. PMID 25646323